CLINICAL TRIAL: NCT04559529
Title: Pharmacological Modulation of Hippocampal Activity in Psychosis 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Stephan Heckers, Dept Chairperson Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: VEPP_200915
Record Dates: First submitted 2020-09-16; First posted 2020-09-23 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Levetiracetam; Levamisole

STUDY DESIGN:
Intervention Model Description: 2-way crossover, double-blind, randomized controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: During Visit 2, participants will be randomly assigned to an intervention arm in which they will receive two 250mg LEV capsules or two placebo capsules. Both the participant and the research team will be blinded to which arm each participant is in. During Visit 3, the participant will undergo cross-over and receive either two 250mg LEV capsules or two placebo capsules (whichever intervention they did not receive in Visit 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Levetiracetam (LEV), then Placebo (Experimental): Participants will first receive two 250mg LEV capsules on the same day. After one week, they will receive two placebo capsules on the same day.
  Interventions: Drug: Levetiracetam (LEV) 500 mg; Drug: Placebo
- Placebo, then Levetiracetam (LEV) (Experimental): Participants will first receive two placebo capsules on the same day. After one week, they will receive two 250mg LEV capsules on the same day.
  Interventions: Drug: Levetiracetam (LEV) 500 mg; Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam (LEV) 500 mg — The levetiracetam pill will look just like the placebo pill.
  Other Names: Keppra
Drug: Placebo — The placebo pill will look just like the levetiracetam pill, but does not contain any levetiracetam.

SUMMARY:
The purpose of this study is to test whether administration of levetiracetam (LEV), a commonly used anti-epileptic that alters neurotransmitter release, can reduce hippocampal hyperactivity in people with psychotic disorders. Specifically, the investigators will utilize two functional magnetic resonance imaging (MRI) techniques: 1) blood-oxygen-level-dependent (BOLD) contrast will assess activity with a visual scene processing task that engages the anterior hippocampus and 2) arterial spin labeling (ASL) will assess baseline activity. Previous studies in people with psychotic disorders have shown that the hippocampus is hyperactive and more activity correlates with worsening of clinical symptoms. Therefore, the aim of this study is to use an intervention to further understand the underlying mechanisms of the hippocampus in psychosis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for psychosis subjects

1. Men and women age 18 - 65.
2. Communicative in English.
3. Provide voluntary, written informed consent.
4. Physically healthy by medical history.
5. BMI > 17.5 and < 45.
6. Diagnosis of a psychotic disorder confirmed by Structured Clinical Interview for Diagnostic and Statistical Manual-5 (SCID) or diagnostic interview with a trained clinician.
7. Stable medication regimen over at least the past two weeks, including the use of either an oral or intramuscular administration of an antipsychotic medication.
8. For females, no longer of child-bearing potential, or agreeing to practice effective contraception during the study (e.g., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; barrier methods: condom with spermicidal foam/gel/film/cream/suppository or occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam/gel/film/cream/suppository; male partner sterilization; or true abstinence when this is in line with the preferred and usual lifestyle of the subject); and,
9. For females of child-bearing potential, must have a negative urine pregnancy test before MRI and drug administration.
10. Not breastfeeding/nursing at time of screening or at any time during the study.

Inclusion criteria for healthy controls

1. All of the above except for subjects will be psychiatrically healthy and not taking psychotropic or potentially psychoactive prescription medication.

----

Exclusion Criteria:

Exclusion criteria for psychosis subjects

1. Age less than 18 or greater than 65.
2. Not communicative in English.
3. Unable to provide written informed consent.
4. Current medical or neurological illness.
5. History of severe head trauma.
6. BMI < 17.5 or > 45.
7. Meets criteria for diagnosis of substance or alcohol use disorder within the past month.
8. Positive urine pregnancy test during the study.
9. Breastfeeding/nursing at time of screening or at any time during the study.
10. Conditions that preclude MR scanning (as defined in the Screening Form)
11. Conditions that preclude study drug administration (as defined in the Screening Form)

Exclusion criteria for healthy controls

All of the above and in addition:

1. Current use of psychotropic or potentially psychoactive prescription medication.
2. Major psychiatric disorder as determined by Diagnostic and Statistical Manual -5 (major depression, bipolar disorder, obsessive compulsive disorder, post-traumatic stress disorder, etc)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Heckers, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Control Participants: Levetiracetam (LEV), Then Placebo: Healthy control participants will first receive two 250mg LEV capsules on the same day. After one week, they will receive two placebo capsules on the same day.
- Healthy Control Participants: Placebo, Then Levetiracetam (LEV): Healthy control participants will first receive two placebo capsules on the same day. After one week, they will receive two 250mg LEV capsules on the same day.
- Patients With Schizophrenia: Levetiracetam (LEV), Then Placebo: Participants with schizophrenia will first receive two 250mg LEV capsules on the same day. After one week, they will receive two placebo capsules on the same day.
- Patients With Schizophrenia: Placebo, Then Levetiracetam (LEV): Participants with schizophrenia will first receive two placebo capsules on the same day. After one week, they will receive two 250mg LEV capsules on the same day.
Period: First Intervention (1 Day)
Arm/Group | Healthy Control Participants: Levetiracetam (LEV), Then Placebo | Healthy Control Participants: Placebo, Then Levetiracetam (LEV) | Patients With Schizophrenia: Levetiracetam (LEV), Then Placebo | Patients With Schizophrenia: Placebo, Then Levetiracetam (LEV)
Started | 15 | 15 | 15 | 17
Completed | 15 | 15 | 14 | 16
Not Completed | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawn due to inability to complete imaging | 0 | 0 | 1 | 0
Period: Washout (At Least 7 Days)
Arm/Group | Healthy Control Participants: Levetiracetam (LEV), Then Placebo | Healthy Control Participants: Placebo, Then Levetiracetam (LEV) | Patients With Schizophrenia: Levetiracetam (LEV), Then Placebo | Patients With Schizophrenia: Placebo, Then Levetiracetam (LEV)
Started | 15 | 15 | 14 | 16
Completed | 15 | 15 | 14 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Healthy Control Participants: Levetiracetam (LEV), Then Placebo | Healthy Control Participants: Placebo, Then Levetiracetam (LEV) | Patients With Schizophrenia: Levetiracetam (LEV), Then Placebo | Patients With Schizophrenia: Placebo, Then Levetiracetam (LEV)
Started | 15 | 15 | 14 | 16
Completed | 15 | 15 | 13 | 16
Not Completed | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Control Participants: Levetiracetam (LEV), Then Placebo: Healthy control participants will undergo two MRI scanning sessions. Each session includes two functional magnetic resonance imaging (MRI) techniques:
  1. Blood-oxygen-level-dependent (BOLD) contrast to assess activity with a visual scene processing task that engages the hippocampus.
  2. Arterial spin labeling (ASL) to assess baseline activity. ASL measures cerebral blood flow, which is linked to neuronal metabolism and functions as a proxy for neuronal activity.
  About 2 hours before the first imaging session, they will receive levetiracetam (LEV) 500 mg. The levetiracetam pill will look just like the placebo pill. About 2 hours before the second imaging session, they will receive the placebo pill. The placebo pill will look just like the levetiracetam pill, but does not contain any levetiracetam.
- Healthy Control Participants: Placebo, Then Levetiracetam (LEV): Healthy control participants will undergo two MRI scanning sessions. Each session includes two functional magnetic resonance imaging (MRI) techniques:
  1. Blood-oxygen-level-dependent (BOLD) contrast to assess activity with a visual scene processing task that engages the hippocampus.
  2. Arterial spin labeling (ASL) to assess baseline activity. ASL measures cerebral blood flow, which is linked to neuronal metabolism and functions as a proxy for neuronal activity.
  About 2 hours before the first imaging session, they will receive the placebo pill. The placebo pill will look just like the levetiracetam pill, but does not contain any levetiracetam. About 2 hours before the second imaging session, they will receive levetiracetam (LEV) 500 mg. The levetiracetam pill will look just like the placebo pill.
- Patients With Schizophrenia: Levetiracetam (LEV), Then Placebo: Patients with schizophrenia will undergo two MRI scanning sessions. Each session includes two functional magnetic resonance imaging (MRI) techniques:
  1. Blood-oxygen-level-dependent (BOLD) contrast to assess activity with a visual scene processing task that engages the hippocampus.
  2. Arterial spin labeling (ASL) to assess baseline activity. ASL measures cerebral blood flow, which is linked to neuronal metabolism and functions as a proxy for neuronal activity.
  About 2 hours before the first imaging session, they will receive levetiracetam (LEV) 500 mg. The levetiracetam pill will look just like the placebo pill. About 2 hours before the second imaging session, they will receive the placebo pill. The placebo pill will look just like the levetiracetam pill, but does not contain any levetiracetam.
- Patients With Schizophrenia: Placebo, Then Levetiracetam (LEV): Patients with schizophrenia will undergo two MRI scanning sessions. Each session includes two functional magnetic resonance imaging (MRI) techniques:
  1. Blood-oxygen-level-dependent (BOLD) contrast to assess activity with a visual scene processing task that engages the hippocampus.
  2. Arterial spin labeling (ASL) to assess baseline activity. ASL measures cerebral blood flow, which is linked to neuronal metabolism and functions as a proxy for neuronal activity.
  About 2 hours before the first imaging session, they will receive the placebo pill. The placebo pill will look just like the levetiracetam pill, but does not contain any levetiracetam. About 2 hours before the second imaging session, they will receive levetiracetam (LEV) 500 mg. The levetiracetam pill will look just like the placebo pill.
- Total: Total of all reporting groups
Arm/Group | Healthy Control Participants: Levetiracetam (LEV), Then Placebo | Healthy Control Participants: Placebo, Then Levetiracetam (LEV) | Patients With Schizophrenia: Levetiracetam (LEV), Then Placebo | Patients With Schizophrenia: Placebo, Then Levetiracetam (LEV) | Total
Number analyzed (Participants) | 15 | 15 | 14 | 16 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (9.0) | 36.0 (11.2) | 35.7 (12.1) | 34.8 (12.7) | 34.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 5 | 4 | 18
  Male | 10 | 11 | 9 | 12 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 1 | 4
  Not Hispanic or Latino | 12 | 15 | 14 | 15 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 0 | 6 | 13
  White | 12 | 8 | 14 | 10 | 44
  More than one race | 0 | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 14 | 16 | 60

OUTCOME MEASURES:

1. Primary Outcome: Hippocampal Activity (Arterial Spin Labeling [ASL] Study) After Levetiracetam (LEV)
Description: ASL signal after LEV, using Magnetic Resonance Imaging (MRI) scanning of the brain. ASL measures cerebral blood flow, which is linked to neuronal metabolism and functions as a proxy for neuronal activity.
Time Frame: 2 hours after LEV administration
Population: The overall number of participants analyzed is inconsistent with the numbers provided in the participant flow module due to MRI scanner or participant error during the collection of the ASL sequence. However, these participants still included useful imaging data collected in other imaging sequences during the study.
Measure: Mean (95% Confidence Interval); unit: ml/100g/min
Arm/Group | Healthy Control Participants: Levetiracetam (LEV), Then Placebo | Healthy Control Participants: Placebo, Then Levetiracetam (LEV) | Patients With Schizophrenia: Levetiracetam (LEV), Then Placebo | Patients With Schizophrenia: Placebo, Then Levetiracetam (LEV)
Number analyzed (Participants) | 15 | 14 | 14 | 14
ml/100g/min | 28.3 [25.2 to 31.3] | 27.1 [24.9 to 29.4] | 28.0 [24.7 to 31.3] | 28.5 [25.5 to 31.5]

2. Primary Outcome: Hippocampal Activity (Arterial Spin Labeling [ASL] Study) After Placebo
Description: ASL signal after placebo, using Magnetic Resonance Imaging (MRI) scanning of the brain. ASL measures cerebral blood flow, which is linked to neuronal metabolism and functions as a proxy for neuronal activity.
Time Frame: 2 hours after placebo administration
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ml/100g/min
Arm/Group | Healthy Control Participants: Levetiracetam (LEV), Then Placebo | Healthy Control Participants: Placebo, Then Levetiracetam (LEV) | Patients With Schizophrenia: Levetiracetam (LEV), Then Placebo | Patients With Schizophrenia: Placebo, Then Levetiracetam (LEV)
Number analyzed (Participants) | 13 | 15 | 13 | 14
ml/100g/min | 28.1 [25.6 to 30.5] | 28.3 [25.2 to 31.4] | 28.1 [25.5 to 30.7] | 28.7 [25.5 to 32.0]

3. Primary Outcome: Hippocampal Recruitment (Blood-Oxygen-Level-Dependent [BOLD] Study) After Levetiracetam (LEV)
Description: BOLD signal after LEV, using Magnetic Resonance Imaging (MRI) scanning of the brain. This method reflects changes in oxygenation of blood in the brain during a scene-processing task that engages, or recruits, the hippocampus.
Time Frame: 2 hours after LEV administration
Population: The overall number of participants analyzed is inconsistent with the numbers provided in the participant flow module due to MRI scanner or participant error during the collection of the recruitment data using the BOLD signal. However, these participants still included useful imaging data collected in other imaging sequences during the study.
Measure: Mean (95% Confidence Interval); unit: BOLD percent signal change
Arm/Group | Healthy Control Participants: Levetiracetam (LEV), Then Placebo | Healthy Control Participants: Placebo, Then Levetiracetam (LEV) | Patients With Schizophrenia: Levetiracetam (LEV), Then Placebo | Patients With Schizophrenia: Placebo, Then Levetiracetam (LEV)
Number analyzed (Participants) | 15 | 14 | 13 | 11
BOLD percent signal change | -0.0342 [-0.2172 to 0.1489] | 0.1216 [-0.0382 to 0.2813] | 0.2915 [0.1084 to 0.4745] | 0.2381 [-0.0078 to 0.4840]

4. Primary Outcome: Hippocampal Recruitment (Blood-Oxygen-Level-Dependent [BOLD] Study) After Placebo
Description: BOLD signal after placebo, using Magnetic Resonance Imaging (MRI) scanning of the brain. This method reflects changes in oxygenation of blood in the brain during a scene-processing task that engages, or recruits, the hippocampus.
Time Frame: 2 hours after placebo administration
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: BOLD percent signal change
Arm/Group | Healthy Control Participants: Levetiracetam (LEV), Then Placebo | Healthy Control Participants: Placebo, Then Levetiracetam (LEV) | Patients With Schizophrenia: Levetiracetam (LEV), Then Placebo | Patients With Schizophrenia: Placebo, Then Levetiracetam (LEV)
Number analyzed (Participants) | 14 | 14 | 12 | 14
BOLD percent signal change | 0.1908 [-0.0158 to 0.3975] | 0.0507 [-0.1081 to 0.2094] | 0.1769 [-0.0607 to 0.4146] | 0.0703 [-0.1121 to 0.2526]

ADVERSE EVENTS:
Time Frame: Up to 4 hours after levetiracetam or placebo administration.
Groups:
- Healthy Control Participants: Levetiracetam (LEV): All healthy control participants that received LEV. All individuals contributed data to the study outcomes.
- Healthy Control Participants: Placebo: All healthy control participants that received placebo. All individuals contributed data to the study outcomes.
- Patients With Schizophrenia: Levetiracetam (LEV): All patients with schizophrenia that received LEV, including individuals that did not contribute data to the study outcomes.
- Patients With Schizophrenia: Placebo: All patients with schizophrenia that received placebo, including individuals that did not contribute data to the study outcomes.
Arm/Group | Healthy Control Participants: Levetiracetam (LEV) | Healthy Control Participants: Placebo | Patients With Schizophrenia: Levetiracetam (LEV) | Patients With Schizophrenia: Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/31 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Control Participants: Levetiracetam (LEV) (N=30) | Healthy Control Participants: Placebo (N=30) | Patients With Schizophrenia: Levetiracetam (LEV) (N=31) | Patients With Schizophrenia: Placebo (N=30)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT04559529/Prot_SAP_000.pdf